CLINICAL TRIAL: NCT01631344
Title: Intervention Study to Examine the Effectiveness of Lifestyle Counseling Using the "Stage of Change" Model Versus Conventional Physical Therapy on Chronic Low Back Pain
Brief Title: Effectiveness of Lifestyle Counseling Versus Physical Therapy on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008036
Record Dates: First submitted 2012-06-07; First posted 2012-06-29 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Therapy (No Intervention): Conventional Physical Therapy
- Daily physical activity consultation, Using Stage of change (Experimental)
  Interventions: Other: Daily physical activity consultation, Using the "Stage of change" model

INTERVENTIONS:
Other: Daily physical activity consultation, Using the "Stage of change" model — Consultation of daily physical activity is provided, including selection of up to four pain relief exercises
  Arms: Daily physical activity consultation, Using Stage of change

SUMMARY:
Background:

Low back pain is the leading cause of disability, affecting the quality of life and work productivity.

It is the most common reason for seek medical help and advice. Low back pain creates huge economical burden worldwide. To date, most ( 90%) of low back pain cases are not clinically defined with no preferred medical treatment

1. Study objectives:

   To prove that consulting using the "Stage of change" model for daily physical activity will lead to long term improvement of pain, disability and well-being parameters of those suffering from chronic low back pain, people age 25-55, when compared to conventional Physical Therapy.
2. Study hypotheses:

   The intervention groups vs. Physical Therapy group will demonstrate that the following parameters will improve after: 3 months, one, two and five years.
   1. Pain reduction.
   2. Less disability - improvement in daily activities.
   3. Better feeling of health and well-being.
   4. Increased and better compliance to daily sport activities.
   5. BMI reduction.
   6. Reduction of cigarette smoking.
   7. Reduction of usage of anti-analgesics and anti-inflammatory medications.
   8. Reduction in number of visits to Physical Therapy clinics due to low back pain.
3. Methods:

The present Randomized intervention study that will include 220 healthy individuals, males and females aged 25-55 years old suffering from chronic or recurrent low back pain, with or without radiation to the legs that were referred to Maccabi Healthcare Services Physical Therapy clinics in the Sharon district in Israel.

These individuals will be randomized to one of the following two groups:

1. Conventional Physical Therapy.
2. Physical Therapy focused on healthy lifestyle using the "Stage of Change" model.

Non-dependent observer will follow-up on the outcome parameters via phone calls and filling the questionnaire's with the relevant study participants following 3 months, 1 year, 2 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 25-55 years old
* Chronic / recurrent low back pain (over 3 months)
* With or without radiation

Exclusion Criteria:

* Rheumatoid disease
* Tumors
* Fibromyalgia
* Back surgery
* Road / work accidents
* Non Hebrew speaking
* Pregnancy

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2011-02; Primary Completion 2017-07 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Disability using the Roland Morris Disability Questionnaire at 3 months, 1, 2 and 5 years | 3 months, 1, 2 and 5 years

SECONDARY OUTCOMES:
Change from baseline of Pain using the Numerical pain scale at 3 months, 1, 2 and 5 years | 3 months, 1, 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yair Shapiro, MD., Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Maccabi Healthcare Services Clinics, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Canaway A, Pincus T, Underwood M, Shapiro Y, Chodick G, Ben-Ami N. Is an enhanced behaviour change intervention cost-effective compared with physiotherapy for patients with chronic low back pain? Results from a multicentre trial in Israel. BMJ Open. 2018 Apr 10;8(4):e019928. doi: 10.1136/bmjopen-2017-019928. PMID 29643158
- [Derived] Ben-Ami N, Shapiro Y, Pincus T. Outcomes in Distressed Patients With Chronic Low Back Pain: Subgroup Analysis of a Clinical Trial. J Orthop Sports Phys Ther. 2018 Jun;48(6):491-495. doi: 10.2519/jospt.2018.7670. Epub 2018 Mar 27. PMID 29587572
- [Derived] Ben-Ami N, Chodick G, Mirovsky Y, Pincus T, Shapiro Y. Increasing Recreational Physical Activity in Patients With Chronic Low Back Pain: A Pragmatic Controlled Clinical Trial. J Orthop Sports Phys Ther. 2017 Feb;47(2):57-66. doi: 10.2519/jospt.2017.7057. PMID 28142364